CLINICAL TRIAL: NCT00339157
Title: ANAkinra in Severe Juvenile Idiopathic Arthritis of Systemic Onset (ANAJIS)
Brief Title: Interleukin-1 Receptor Antagonist (IL-1RA) (ANAKINRA) IN SEVERE SYSTEMIC-ONSET JUVENILE IDIOPATHIC ARTHRITIS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C05-40
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Systemic-Onset Juvenile Idiopathic Arthritis
Keywords: IDIOPATHIC JUVENILE ARTHRITIS; PEDIATRICS; ORPHAN DISEASE; INTERLEUKIN - 1; RECEPTORS , INTERLEUKINS; ANTAGONISTS
MeSH Terms: conditions — Arthritis, Juvenile; Rare Diseases | interventions — Interleukin 1 Receptor Antagonist Protein; Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Anakinra
Biological: Pneumo23

SUMMARY:
1. Main objective: To test the efficacy of anakinra treatment in children or young adults with corticosteroid-resistant or -dependent Systemic-Onset Juvenile Idiopathic Arthritis (SO-JIA)
2. Design: Double blind, randomized trial testing the efficacy of one month Anakinra treatment versus placebo (2 groups of 12 patients each). All the patients will be treated with anakinra during the following 11 months and the dose of corticosteroids will be gradually tapered (= descriptive part of the trial to assess the tolerance and efficacy over 12 months).
3. Hypothesis: 70% significant improvement after 1 month in Anakinra-treated patients versus no more than 10% in the placebo group.
4. Main inclusion criteria : diagnosis of SO-JIA (Durban consensus conference criteria), age: 2 to 20 years at inclusion, active, corticosteroid-resistant or -dependent disease, no previous IL-1ra treatment.

ELIGIBILITY:
Inclusion Criteria:

* SO-JIA (Edmonton's revision of Durban's consensus conference criteria)
* Age: at least 2 years and less than 20 years at treatment initiation
* Disease duration of at least 6 months
* Failure of corticosteroid treatment or requirement for corticosteroid treatment at a daily dose equal to or over 0.3 mg/kg (10 mg in patients whose weight is over 34 kg)
* Active and severe systemic symptoms and/or arthritis as assessed by an experienced pediatric Rheumatologists, with at least 3 of the following criteria when assessing Giannini's core-set items: 1) physician global assessment of disease activity of at least 20/100; 2) parent/patient assessment of disease effect on overall well-being of at least 20/100; 3) functional disability with a Children Health Assessment Questionnaire (CHAQ, Ref [9]) score equal to or higher than 0.375/3; 4) 2 joints or more with active arthritis 5) 2 joints or more with non-irreversible limited range of motion (irreversible limited range of motion will be defined by radiological evidence of irreversible joint damage and ankylosis) 6) erythrocyte sedimentation rate (ESR) equal to or higher than 20.
* In the absence of disease-related fever, either CRP or first hour ESR or both have to be over the upper limit of normal values so that treatment effect on the systemic part of the disease can be objectively evaluated.
* Patients with polyarthritis (at least 5 joints with inflammation and/or limitation of motion) will be eligible for this study only if at least 50% of the affected joints do not present radiological evidence of irreversible damage.
* Informed consent signed by the parents or the person legally responsible for the patient if the patient is less than 18, and by the patient if old enough
* Teenager girls or young women with childbearing potential must use a contraceptive method (including abstinence
* tuberculin test performed before Day 1 and must either be negative or positivity must be related to previous immunization and of normal intensity according to the investigator's judgment

Exclusion Criteria:

* Previous treatment with IL-1Ra
* intra-articular injection or change in the doses of non-steroidal anti-inflammatory drugs and corticosteroids in the 4 weeks preceding the initiation of anakinra treatment
* Treatment with another immunosuppressive or disease-modifying drugs that could not be stopped before inclusion (for a duration depending on the drug pharmacokinetic properties)
* Contra-indication to the use of anakinra including ongoing active infection or allergy to E Coli's derivate or other components of the drug
* Previous history of malignancy or heart insufficiency
* Patients with asthma require to be previously assessed by a pneumonologist
* Obvious need of therapeutic intervention before study completion such as surgery, intra-articular injection, life vaccine administration
* Any of the following: leucocyte counts < 3.6 x 10e9/L, polymorphonuclear neutrophil counts < 1.5 x 10e9/L, platelets < 150 000/mm3, serum creatinin > 1.5 the upper limit of normal range for age, serum alanine and aspartate transaminases > 2 times the upper limit of the normal range, serum bilirubin > 2 times the upper limit of the normal range

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24
Dates: Start 2006-06; Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
30% improvement of JIA activity after 1 month compared to day 1 according to Giannini's core-set criteria, ie 30% improvement of at least 3 of the 6 items and no more than one item worsened by 30% or more.
Number of active arthritis
Number of joints with limitation of motion
Physician assessment of disease activity
Parent or patient's assessment of disease activity
Childhood health assessment questionnaire
First hour ESR)
Improvement of systemic symptoms between day 1 and month 1 as assessed by the resolution of the fever if present initially, by a 50% decrease or a normalization of the C-reactive protein and of the first hour ES

SECONDARY OUTCOMES:
Number, severity and type of adverse events over 12 months
Proportion of patients reaching 50%, 70% and 100% improvement of JIA activity according to Giannini's core-set criteria at each visit (day 15, month 1 to 6, month 9 and month 12)
Proportion of patients in whom the daily dose of corticosteroids can be reduced to less than 0.3 mg/kg (less than 10 mg in patients over 34 kg) at month 6
Proportion of patients with a normalization of the glycosylated ferritin / ferritin ratio (if lower than 1/4 initially) after 1, 2 and 6 months
Variation of cytokine expression by PBMC between Day 1 and Month 1 and Month 6
Antibody response at month 1 and month 6 to Pneumo 23® immunization: immunization on day 1 against Streptococcus pneumoniae
Pharmacokinetic study at month 2 and month 6

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Quartier-dit-Maire, MD, Principal Investigator — Pediatric Immuno-Hematology and Rheumatology Unit, Necker-Enfants Malades Hospital, 149 rue de Sevre, 75015 Paris, France
Locations (6):
- France (6):
  - Bordeaux CHU, Bordeaux
  - Kremlin-Bicetre Hospital, Le Kremlin-Bicêtre
  - Hopital Lyon Edouard Herriot, Lyon
  - Nancy Hopital d'Enfants, Nancy
  - Pediatric Immuno-Hematology and Rheumatology Unit, Necker-Enfants Malades Hospital, 149 rue de Sevres, Paris
  - Robert Debre Hospital, Paris

REFERENCES:
- [Derived] Quartier P, Allantaz F, Cimaz R, Pillet P, Messiaen C, Bardin C, Bossuyt X, Boutten A, Bienvenu J, Duquesne A, Richer O, Chaussabel D, Mogenet A, Banchereau J, Treluyer JM, Landais P, Pascual V. A multicentre, randomised, double-blind, placebo-controlled trial with the interleukin-1 receptor antagonist anakinra in patients with systemic-onset juvenile idiopathic arthritis (ANAJIS trial). Ann Rheum Dis. 2011 May;70(5):747-54. doi: 10.1136/ard.2010.134254. Epub 2010 Dec 20. PMID 21173013